CLINICAL TRIAL: NCT02553473
Title: Six Versus Two Weeks Treatment With Doxycycline in Lyme Neuroborreliosis; a Multicenter, Non-inferiority, Penta-blind, Randomized Trial
Brief Title: Six Versus Two Weeks Treatment With Doxycycline in Lyme Neuroborreliosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-001481-25
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2021-06

CONDITIONS: Neuroborreliosis, Borrelia Burgdorferi
MeSH Terms: conditions — Lyme Neuroborreliosis | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Doxycycline for 6 weeks (Active Comparator): Doxycycline 200 mg once daily for six weeks
  Interventions: Drug: Doxycycline
- Doxycycline for 2 weeks + placebo (Placebo Comparator): Doxycycline 200 mg once daily for two weeks + placebo for four weeks.
  Interventions: Drug: Doxycycline; Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline
Drug: Placebo
  Arms: Doxycycline for 2 weeks + placebo

SUMMARY:
Comparison of Doxycycline 200 mg once daily for six weeks versus Doxycycline 200 mg once daily for two weeks + placebo for four weeks. Primary objective is to answer the question "is two weeks doxycycline treatment (currently suggested treatment) at least as effective as six weeks doxycycline treatment in Lyme Neuroborreliosis?".Key secondary objectives are to provide a better understanding of the pathogenesis and long-term complaints, and to search for new biomarkers in Lyme Neuroborreliosis (LNB) by collecting clinical data, blood, and cerebrospinal fluid (CSF) in a biobank for future research

Endpoints:

Primary endpoint: Improvement on a composite clinical score from inclusion to six months after ended treatment defined as clinical score at inclusion minus clinical score at six months.

Secondary endpoints: Improvement on a composite clinical score 12 months after ended treatment. Fatigue Severity Scale (FSS),Patient Health Questionnaire (PHQ-15), Short Form 36 (SF-36) and blood and CSF findings at inclusion, after 6 and 12 months.

The study design is a multicenter, non-inferiority, randomized, penta-blind, placebo-controlled trial. 120 patients will be included from approximately 8 Norwegian hospitals.

Main inclusion criteria are neurological symptoms suggestive of LNB without other obvious reasons, one or both of a) Cerebrospinal fluid pleocytosis (>5 leukocytes/mm3) b) intrathecal Bb antibody Production and signed informed consent. Safety assessments during the trial: Comparison of clinical outcome six months after end of treatment between the two treatment groups. Subjective experiences and blood tests including hematology and biochemistry for four weeks after ended treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Neurological symptoms suggestive of LNB without other obvious reasons and one or both of

   1. Cerebrospinal fluid pleocytosis ≥5 leukocytes pr mm3
   2. Intrathecal Bb antibody production
2. Signed informed consent

Exclusion Criteria:

* Age less than 18 years
* Pregnancy, breast-feeding
* Adverse reaction to tetracyclines
* Treatment with cephalosporin, penicillin, or tetracycline the last 14 days
* Serious liver or kidney disease that contraindicates use of doxycycline
* Lactose intolerance
* Need to use medications contraindicated according to Summary of Product Characteristics of the Investigational Medicinal Product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marit Solheim, M.D, Principal Investigator — Sørlandet hospital HF

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline for 6 Weeks: Doxycycline 200 mg once daily for six weeks
  Doxycycline
- Doxycycline for 2 Weeks + Placebo: Doxycycline 200 mg once daily for two weeks + placebo for four weeks.
  Doxycycline
  Placebo
Period: Overall Study
Arm/Group | Doxycycline for 6 Weeks | Doxycycline for 2 Weeks + Placebo
Started | 61 | 60
Completed | 54 | 55
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline for 6 Weeks | Doxycycline for 2 Weeks + Placebo | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15) | 58 (12) | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 32 | 35 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 61 | 60 | 121
Region of Enrollment [Count of Participants; unit: Participants]
  Norway | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Difference in Composite Clinical Score From Inclusion to Six Months After Ended Treatment
Description: Clinical change on composite clinical score (CCS) defined as score at inclusion minus score at 6 months after treatment.CCS consisted of 32 variables,scored from 0 to 2 points.Minimum 0 points,maximum 64 points.High scale score indicated worse outcome.
  Variables scored:Malaise,Fatigue,Headache,Neck and/or back pain,Abdominal and/or breast pain,Arm pain,Leg pain,Generalised pain located to joints and/or muscles,Memory and/or concentration problems,Other,Facial palsy,Paresis of the eye muscles,Reduced hearing,Other cranial neuropathies,Cervical radicular sensory findings,Cervical radicular paresis,Thoracic radicular sensory findings,Lumbar radicular sensory findings,Lumbar radicular paresis,Non-radicular sensory findings,Non-radicular paresis,Other,Central findings in one extremity,Central findings in a hemi pattern,Central findings in both legs,Central findings in all extremities,Gait ataxia,Dysphasia/aphasia, Nystagmus,Involuntary movement including tremor,Cognitive impairment,Other.
Time Frame: Six months after end of treatment.
Population: Intention to treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Doxycycline for 6 Weeks | Doxycycline for 2 Weeks + Placebo
Number analyzed (Participants) | 53 | 52
units on a scale | 6.4 [5.6 to 7.2] | 6.4 [5.5 to 7.2]

ADVERSE EVENTS:
Time Frame: Follow-up period of 12 months. Patient diary filled out for 10 weeks after start of treatment. Blood sampling at 2 and 4 weeks after start of treatment.
Description: Definition used from Good Clinical Practice. In addition registered patient reported symptoms of side effects.
Arm/Group | Doxycycline for 6 Weeks | Doxycycline for 2 Weeks + Placebo
All-Cause Mortality (participants affected / at risk) | 1/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT02553473/Prot_SAP_000.pdf